CLINICAL TRIAL: NCT06719154
Title: Prospective, Multicentric, Controlled, Double Arm Clinical Investigation to Evaluate the Safety and Efficacy of Profhilo® Structura for Face Adipose Tissue Restoration
Brief Title: Evaluation of the Safety and Efficacy of Profhilo® Structura
Status: Recruiting | Type: Observational
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry); IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 23E3318
Record Dates: First submitted 2024-04-17; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Skin Aging
Keywords: aging; adipose tissue
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treated group: 120 subjects will be treated
  Healthy subjects Male and Female subjects. Age : between 35 and 55 year
  Interventions: Device: Profhilo Structura
- Not treated group: 44 subjects will be not treated
  Healthy subjects Male and Female subjects. Age : between 35 and 55 year
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Device: Profhilo Structura — 2 injections (30 days apart) of investigated medical device into superficial fat compartments of zygomatic arch and preauricular area
  Groups: Treated group
Other: Sham (No Treatment) — Sham (No Treatment)
  Groups: Not treated group

SUMMARY:
Profhilo® Structura is composed of a buffered saline solution of high molecular weight (H-HA) and low molecular weight (L-HA) hyaluronic acid. The high- and low-molecular-weight HA used in the device is obtained by biofermentation and has not undergone chemical modification processes; this results in excellent tolerability of the product.

In addition, the HA chains with different molecular weight present in Profhilo® Structura, thanks to a specific and patented treatment of the solution (NAHYCO® Hybrid Technology), interact with each other, giving Profhilo® Structura unique rheological properties that allow higher concentrations of HA to be administered at equal viscosity of the solution.

The formulation based on HA with different molecular weight contained in Profhilo® Structura is based on the Hydrolift® Action system, the innovative approach aimed at combating the physiological decrease of HA in the skin, restoring hydration, elasticity and tone, synergistically associating deep hydration with the mechanical lifting action of the skin depression.

Thanks to its rheological properties and cohesivity Profhilo® Structura is able to optimally spread and integrate into the interstitial spaces of the adipose tissue. Profhilo® Structura has the specific indication for adipose tissue restoration and is able to counteract facial volume loss.

DETAILED DESCRIPTION:
Profhilo® Structura (HILOW 4.5% hyaluronic acid [HA] sodium salt for intradermal use; developed by IBSA Farmaceutici Italia Srl) is the first Conformité Européenne (CE)-certified HA-based injectable, sterilized, apyrogenic, and resorbable product indicated for female or male adults with mild-to-moderate volume loss in the face or neck to restore adipose tissue, correct and fill natural and induced cutaneous depressions, and improve skin laxity. Profhilo® Structura is also indicated for dermal tissue repair in adults with acne scars.

Profhilo® Structura contains a combination of high and low molecular weight HA chains that interact with each other for unique rheological characteristics that enable the administration of higher concentrations of HA, without an increase in viscosity.

Profhilo® Structura has a corrective/filling action on natural and induced skin depressions formed because of reduced endogenous HA levels and skin hydration, alteration of elastic fibers and collagen in the dermis, and loss of turgor and skin tone (all characteristics which can occur following excessive dehydration, weight loss, or aging). Administered subcutaneously by qualified personnel, the viscoelastic and moisturizing properties of the HA in Profhilo® Structura and the ability to maintain HA to adequate levels within skin tissues using this medical device, enables tissue rehydration, creates optimal conditions for tissue remodeling, and intervenes with the physiological process of skin ageing.

The administration of Profhilo® Structura allows the tissue restoration using the physiological amount of HA. Furthermore, HCC of high and low molecular weight HA combines the regenerating trophic effect of low molecular weight HA on the epidermis (a HYDRO effect), and the plastic modelling effect of high molecular weight HA on the dermis (a LIFT effect, also known as Hydrolift® Action).

Because of its rheological properties and cohesivity, Profhilo® Structura is able to optimally spread and integrate into the interstitial spaces of the adipose tissue. Profhilo® Structura is specifically indicated for adipose tissue restoration and is able to counteract facial volume loss.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects
2. Male and Female subjects.
3. Age : between 35 and 55 year
4. Subject having given freely and expressly his/her informed consent obtained according to ISO 14155:2020 and Good Clinical Practice (GCP)
5. Only for treated group: Subject seeking aesthetic improvement for a corrective/filling action of natural and induced skin depressions
6. Women of childbearing potential must have a negative urine pregnancy test result at inclusion visit and must use a reliable method of contraception since at least 12 weeks and throughout the study.
7. Subject psychologically able to understand the information related to the investigation including possible risks and side effects.
8. Subject able to cooperate with the Investigator and to comply with the requirements of the entire investigation (including ability to attend all the planned investigation visits according to the time limits), based on investigator's judgement.
9. Subject agreeing to keep their usual cleansing / care products during the whole study period.
10. Subject agreeing to apply a SPF50 cream during the whole study period.

Exclusion Criteria:

In terms of population

1. Pregnant or breastfeeding woman or planning a pregnancy during the study.
2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
3. Subject in a social or sanitary establishment.
4. Subject enrolled in another study or whose non-enrollment period is not over.
5. For France only: subject having received a total of 6.000 euros as compensations for their participation in the present study.
6. Subject disagrees to keep a stable weight during the study (BMI variation ± 1)
7. Subject with high expectations for the treatment effect.

   In terms of associated pathology
8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety
9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency
10. Subject suffering from active disease such as inflammation, infection, tumour, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria…) in the 6 months before screening visit
11. Subject with a history of streptococcal disease or an active streptococcus infection
12. Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders.
13. Subject predisposed to keloids or hypertrophic scarring or having healing disorders
14. Subject having history of severe allergy or anaphylactic shock including known risk of hypersensitivity to one of the components of the composition of the investigational device and to antiseptic solution related to previous or current treatment.
15. Subjects with scar, mole, hair or local skin infection (including viral, bacterial, and fungal); skin granulomas; scar constitution; immune system disorders; presence of active or progressive skin disorders or skin diseases with isomorphic response in the treatment area, such as acute eczema, flat wart, lichen planus, psoriasis vulgaris, etc…
16. Patients with psychiatric disorders or emotional instability.

    In terms of previous or ongoing treatment or procedure
17. Any medication which may interfere, at the interpretation of the investigator, with the study objectives.
18. Subject having undergone tooth extraction or dental implant procedure within the past 6 weeks or plans to undergo these procedures during the study.
19. Subject having received facial or cervico-facial lifting in the past 24 months or plans to undergo these procedures during the study.
20. Subject having received treatment with a laser, ultrasound or radiofrequency treatment, a dermabrasion, a surgery, a chemical peeling or any other procedure based on active dermal response on the face within the past 6 months or who plans to undergo any of these procedures during the study.
21. Subject having received within the past 18 months or planning to receive during the study any injections outside of those in the study protocol including non-permanent fillers (e.g., HA, Calcium Hydroxyapatite) or autologous fat on or near the face.
22. Subject having received within the past 9 months or planning to receive during the study any injections outside of those in the study protocol including mesotherapy or botulinum neurotoxin on or near the face.
23. Subject having received at any time or planning to receive a permanent filler on the face (e.g., polylactic acid, Polymethylmethacrylate, silicone) during the study.
24. Subject with subcutaneous retaining structure on the face (meshing, threads, gold strand).
25. Subject having received in the last 24 months resorbable threads lift on the face.
26. Subject having received at any time injection with unknown products
27. Subject using medication such as aspirin, high dose Vitamin C, nonsteroidal anti-inflammatory drugs (NSAIDs), antiplatelet agents, thrombolytics or anticoagulants within one week prior to injection visit or being a chronic user.
28. Subject using medication such as narcotic, and immunosuppressive drugs from three weeks before screening visit and during the whole study period
29. Subject having started or stopped an antidepressant 3 weeks prior the study or plans to use it during the study.
30. Subject undergoing a topical treatment on the face or a systemic treatment:

    * anti-inflammatory medication and/or antihistamines within the past 2 weeks and during the study,
    * corticosteroids within the past 2 weeks and during the study,
    * retinoids and/or immunosuppressors within the past 3 months and during the study.

    In terms of lifestyle
31. Intensive exposure to sunlight or UV-rays within the previous month and/or planning to do so during the study.
32. Heavy smoker (subject who reports smoking 10 or more cigarettes per day);
33. Subject with an excessive consumption of alcohol (more than 2 glasses of wine per day)

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult of both sexes seeking for a corrective/filling action of natural and induced skin depressions.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint | Day 0, Day 30, Day 60, Day 120, Day 180
  Number and percentage of subjects with Adverse Device Effects (ADEs) throughout the study.

SECONDARY OUTCOMES:
Safety endpoint - ISR | Day 0, Day 30, Day 60, Day 120, Day 180
  Number and percentage of subjects with Injection Site Reaction (ISR) and Adverse Events (AEs).
Efficacy endpoint - clinical improvement | Day 0, Day 30, Day 60, Day 120, Day 180
  Percentage of subjects with a clinical improvement from baseline assessed by investigator compared to control group.
Efficacy endpoint - skin quality | Day 0, Day 30, Day 60, Day 120, Day 180
  Percentage of subjects with a skin quality improvement using Beagley-Gibson surface microrelief scale (from grade 1 [Mild] to grade 4 [Severe] from baseline as assessed by investigator compared to control group.
Efficacy endpoint - satisfaction | Day 0, Day 30, Day 60, Day 120, Day 180
  Percentage of positive responders (rated 3 or less) on the GAIS (from grade 1 [Very much improved] to grade 5 [Worse] as assessed by investigator and subjects in live.
Efficacy endpoint - instrumental improvement | Day 0, Day 30, Day 60, Day 120, Day 180
  Percentage of subjects with a instrumental improvement from baseline assessed by investigator compared to control group.

CONTACTS AND LOCATIONS:
Overall Officials: Izabela Błażewicz, MD, Principal Investigator — Eurofins Dermscan Poland
Locations (3):
- Eurofins Dermscan Pharmascan, Villeurbanne, Lyon, France
- Poland (2):
  - Eurofins Dermscan Poland, Gdansk
  - Aesthetic clinical, Poznan

IPD SHARING:
Plan to Share IPD: Undecided